CLINICAL TRIAL: NCT01804647
Title: A One Year Longitudinal Therapeutically Non-Interventional Study of MSRV-Env Burden in Multiple Sclerosis Patients (RRMS - SPMS - PPMS - CIS) as Assessed by PCR and ELISA in Blood
Brief Title: Longitudinal Therapeutically Non-interventional Study of MSRV-Env Burden in Patients With Multiple Sclerosis Disease
Acronym: LOMBARD
Status: Completed | Type: Observational
Sponsor: GeNeuro Innovation SAS (Industry)
Responsible Party: Sponsor
Organization: GeNeuro SA (Industry)
Other Study IDs: GN-E-002
Record Dates: First submitted 2013-03-04; First posted 2013-03-05 (Estimated); Last update posted 2020-10-20 (Actual); Status verified 2018-02

CONDITIONS: Multiple Sclerosis (MS); Relapsing-Remitting MS; Primary Progressive MS; Secondary Progressive MS; Clinically Isolated Syndrome (CIS)
Keywords: Multiple sclerosis (MS); Relapsing-Remitting MS; Primary progressive MS; Secondary progressive MS; Clinically Isolated Syndrome (CIS); Multiple Sclerosis associated RetroVirus (MSRV); MSRV envelop protein (MSRV-Env); Temelimab
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Plasma, serum and PBMC
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- 33 RRMS patients: No study treatments administered
  Interventions: Other: No study treatments administered - blood draws only
- 9 PPMS patients: No study treatments administered
  Interventions: Other: No study treatments administered - blood draws only
- 12 SPMS patients: No study treatments administered
  Interventions: Other: No study treatments administered - blood draws only
- 4 CIS patients: No study treatments administered
  Interventions: Other: No study treatments administered - blood draws only

INTERVENTIONS:
Other: No study treatments administered - blood draws only

SUMMARY:
This study intends to explore evolution of MSRV expression by analyzing the levels of MSRV transcripts in blood, as well as the levels of the MSRV-Env protein in serum of MS patients. The study will be conducted over one year in four cohorts of patients with different forms of MS (remitting-relapsing MS i.e. RRMS, primary-progressive MS i.e. PPMS and secondary-progressive MS i.e. SPMS) and in clinically isolated syndrome (CIS) patients who have suffered a single clinical event but do not comply with diagnosis criteria for definite MS. The MSRV RNA and MSRV-Env protein levels will be correlated with the clinical evolution of patients and with the reverse transcriptase activity, inflammatory markers assessed by cytokines levels. A control group of healthy subjects will be included (the study, GN-E-003, is performed in parallel and is part of another dedicated protocol).

ELIGIBILITY:
Inclusion Criteria:

* Signature of an informed consent;
* Male or female between 18 and 60 years of age;
* Patients with PPMS (Revised McDonald criteria 2010) or patients with SPMS or CIS or patients with RRMS (Revised McDonald criteria 2010) ideally without IFN beta therapy at the T0 visit for RRMS patient only.

Exclusion Criteria:

* Positive serology for hepatitis B or C or HIV;
* Acute infection at inclusion;
* Severe psychiatric disorder;
* Autoimmune disease other than MS;
* Pregnancy or breastfeeding;
* Heavy smokers i.e. more than 10 cigarettes per day;
* History of alcohol or drug abuse in the last 3 years;
* Participation in a clinical trial (within the last 3 months).

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patients coming to the Hospital for regular visits.
Sampling Method: Non-Probability Sample
Enrollment: 58 (Actual)
Dates: Start 2012-11; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Monitor the levels of MSRV-Env expression in MS patients (according to McDonald criteria) of different diagnostic subgroups (RRMS, SPMS, PPMS, CIS) | 1 year
  Monitor the levels of MSRV-Env expression in MS patients (according to McDonald criteria) of different diagnostic subgroups (RRMS, SPMS, PPMS, CIS) over time using 3 approaches:
  * MSRV transcripts in PBMC;
  * MSRV transcripts in plasma;
  * MSRV-Env protein in serum.

SECONDARY OUTCOMES:
Associate the levels of MSRV-Env protein and transcripts | 1 year
Associate the levels of MSRV-Env as assessed with the 3 approaches with MS relapses/exacerbations and/or clinical evolution (EDSS score) and /or treatment | 1 year
Associate the levels of MSRV-Env as assessed with the 3 approaches with levels of inflammatory markers and reverse transcriptase activity | 1 year
Compare levels of MSRV-Env of MS patients to those obtained in a parallel study in Healthy Controls | 1 year

CONTACTS AND LOCATIONS:
Locations (4):
- France (2):
  - Hospices civils de Lyon - Service de Neurologie A - 59 Boulevard Pinel, Bron
  - CHU Timone - Service de Neurologie et CRMBM CNRS 7339 - 264, rue Saint Pierre, Marseille
- Hospital Universitari and Research Institute Vall d'Hebron - Servicio de Neuroimunologia de Nuestro Centro - Pg. Vall d'Hebron 119-129, Barcelona, Catalonia, Spain
- Centre Hospitalier Universitaire Vaudois - Dpt of Clinical Neurosciences - Neurology /Batiment 10-131 - Rue du Bugnon 46 -, Lausanne, Switzerland